CLINICAL TRIAL: NCT07244029
Title: Evaluation of Aescin-Based Herbal Extracts for Managing Postoperative Sequelae Following Impacted Mandibular Third Molar Surgery: A Randomized, Single-Blind, Controlled Trial
Brief Title: Aescin-Based Herbal Extract (Reparil) for Postoperative Sequelae After Mandibular Third Molar Surgery
Acronym: Reparil
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Suhail AlSamari, Principal Investigator - General Dentistry Resident (OMSB), Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCMSS-MREC 030/2025
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Facial Swelling; Trismus
Keywords: Aescin; Escin; Reparil; Ibuprofen; Herbal anti-inflammatory; Postoperative sequelae; Third molar extraction; Oral surgery; Phytotherapeutic agents; Pain management
MeSH Terms: conditions — Pain, Postoperative; Trismus; Agnosia | interventions — Escin; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group, randomized, single-blind controlled clinical trial comparing Reparil (Aescin 20 mg TID) versus Ibuprofen 400 mg TID following surgical extraction of impacted mandibular third molars.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Single-masked: the care provider (surgeon) and the outcomes assessor are blinded to group allocation. Participants are not blinded due to differences in appearance of study medications. Allocation concealment is maintained by coded medication packs prepared by an independent pharmacist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aescin (Reparil®) Group (Experimental): Participants will receive Reparil®-Dragees tablets containing Aescin 20 mg, manufactured by Meda Pharmaceuticals (Germany), administered orally three times daily (TID) for five consecutive days following surgical extraction of an impacted mandibular third molar. A rescue analgesic (Diclofenac potassium 50 mg, Rapidus® by Tabuk Pharmaceutical Manufacturing Co., Saudi Arabia) will be provided if pain is uncontrolled. Clinical assessments will be performed at baseline (preoperatively), on postoperative day 2, and on day 7 for pain (VAS), facial swelling (3D scan), and mouth opening (digital caliper).
  Interventions: Drug: Escin
- Ibuprofen Group (Active Comparator): Participants will receive Ibuprofen tablets 400 mg, manufactured by Flamingo Pharmaceuticals Ltd. (India), administered orally three times daily (TID) for five consecutive days following surgical extraction of an impacted mandibular third molar. Clinical evaluations will be conducted at baseline, postoperative day 2, and day 7 to assess pain intensity (Visual Analog Scale), facial swelling (3D facial scan), and mouth opening (digital caliper).
  Interventions: Drug: Ibuprofen 400 mg

INTERVENTIONS:
Drug: Escin — Oral administration of Aescin 20 mg (Reparil®-Dragees, Meda Pharmaceuticals, Germany), taken three times daily (TID) for five consecutive days following surgical extraction of an impacted mandibular third molar. Each tablet contains 20 mg of purified Aescin derived from Aesculus hippocastanum.
  Other Names: Reparil®-Dragees
  Arms: Aescin (Reparil®) Group
Drug: Ibuprofen 400 mg — Oral administration of Ibuprofen 400 mg tablets (Flamingo Pharmaceuticals Ltd., India), taken three times daily (TID) for five consecutive days following surgical extraction of an impacted mandibular third molar.
  Other Names: Ibuprofen 400 mg Tablets BP
  Arms: Ibuprofen Group

SUMMARY:
This randomized, single-blind, controlled clinical trial aims to evaluate the efficacy and safety of Aescin-based herbal extract (Reparil®) compared with Ibuprofen in managing postoperative sequelae following surgical removal of impacted mandibular third molars. A total of 100 participants aged 18-40 years will be enrolled at the Dental Center, Medical City Hospital for Military and Security Services (MCMSS), Al Khoud, Oman. Participants will be randomly assigned to receive either Reparil® (Aescin 20 mg, three times daily for five days) or Ibuprofen (400 mg, three times daily for five days) following standardized third molar extraction procedures. Postoperative outcomes including pain (VAS), facial swelling (3D facial scanner), and mouth opening (digital caliper) will be assessed preoperatively, on day 2, and day 7 post-surgery. The study aims to determine whether Aescin offers comparable analgesic and anti-edematous effects to Ibuprofen with fewer adverse events.

DETAILED DESCRIPTION:
The extraction of impacted mandibular third molars is one of the most common oral surgical procedures and is frequently associated with pain, facial swelling, and trismus. These postoperative sequelae result from an acute inflammatory response triggered by surgical trauma. Nonsteroidal anti-inflammatory drugs (NSAIDs), particularly Ibuprofen, are widely prescribed for symptom control but are often associated with gastrointestinal, renal, and cardiovascular adverse effects. Hence, safer alternatives with comparable efficacy are being investigated.

Aescin, a natural saponin derived from Aesculus hippocastanum (horse chestnut), exhibits anti-inflammatory, anti-edematous, and venotonic properties. It acts by stabilizing capillary membranes, reducing vascular permeability, and inhibiting the release of inflammatory mediators such as histamine and prostaglandins. Reparil tablets containing Aescin have been clinically validated for treating soft tissue edema and chronic venous insufficiency but have not been extensively evaluated in oral surgical applications.

This prospective, single-center, randomized, single-blind controlled trial will compare the postoperative efficacy of Aescin (Reparil) versus Ibuprofen in patients undergoing surgical extraction of impacted mandibular third molars. Participants will be randomly assigned (1:1) into two treatment groups using computer-generated allocation with pharmacist-controlled concealment. Both the operator and the outcome assessor will be blinded to treatment allocation.

Pain intensity will be measured using a 10-point Visual Analog Scale (VAS). Facial swelling will be objectively assessed using a 3D facial scanner (Revopoint POP 3), and trismus will be measured as the maximum interincisal distance. Assessments will be performed at baseline, postoperative day 2, and day 7. A rescue analgesic (diclofenac sodium 50 mg) will be provided for uncontrolled pain.

All data will be recorded via EpiData version 4.6, with statistical analysis conducted using IBM SPSS Statistics version 30.0. The primary endpoint is postoperative pain reduction; secondary endpoints include facial edema, trismus improvement, and adverse drug effects. This study will contribute to evidence on the use of herbal-based anti-inflammatory agents as potential alternatives to conventional NSAIDs in oral surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for surgical removal of impacted mandibular third molars according to National Institute for Health and Care Excellence (NICE) guidelines.

Age between 18 and 40 years.

Impacted mandibular third molars with similar anatomical position and difficulty level as classified by Pell and Gregory and Pederson scoring.

Healthy individuals (ASA I-II) with no significant systemic illness.

Willing to provide written informed consent and attend all follow-up visits (Day 2 and Day 7 post-surgery).

Exclusion Criteria:

* Recent use (within three weeks preoperatively) of anti-inflammatories, corticosteroids, or antibiotics.

Known allergies or hypersensitivity to Aescin, Ibuprofen, rescue medications, or local anesthetics.

Pregnant or lactating women.

Patients with contraindications to NSAIDs (e.g., asthma, bleeding disorders, chronic kidney disease, active peptic ulcer, or cardiovascular disease).

Recent use of substances that may affect surgery or interact with study drugs (e.g., contraceptives, alcohol, or tobacco).

Surgical time exceeding 30 minutes or cases with intraoperative complications requiring non-study medications.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | Baseline, Day 2, and Day 7 post-surgery
  Change in pain intensity measured using a 10-point Visual Analog Scale (VAS) at baseline (preoperative), postoperative day 2, and postoperative day 7 following surgical extraction of impacted mandibular third molars.

SECONDARY OUTCOMES:
Facial swelling (edema) | Baseline, Day 2, and Day 7 post-surgery
  Change in postoperative facial volume measured using a 3D facial scanner (Revopoint POP 3). Measurements will be taken at baseline (preoperative), postoperative day 2, and postoperative day 7 to assess the degree of facial edema following impacted mandibular third molar surgery.
Mouth opening (trismus) | Baseline, Day 2, and Day 7 post-surgery
  Change in maximum interincisal distance (in millimeters) measured using a digital caliper at baseline (preoperative), postoperative day 2, and postoperative day 7 following surgical extraction of impacted mandibular third molars.
Adverse effects | Baseline to Day 7 post-surgery
  Any drug-related or postoperative adverse effects observed or reported by participants within the 7-day postoperative period will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Suhail H AL Samari, BDS, MFD, Principal Investigator — Oman Medical Speciality Board
Locations (1):
- Medical City for Military and Security Services - Dental Center, Muscat, Al Khoud, Oman

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is a single-center academic clinical trial conducted within a limited institutional setting. Only aggregated and de-identified summary results will be published in peer-reviewed journals and presented at scientific meetings in accordance with institutional and ethical guidelines.

REFERENCES:
- [Background] Bjornsson GA, Haanaes HR, Skoglund LA. Ketoprofen 75 mg qid versus acetaminophen 1000 mg qid for 3 days on swelling, pain, and other postoperative events after third-molar surgery. J Clin Pharmacol. 2003 Mar;43(3):305-14. doi: 10.1177/0091270002250603. PMID 12638400
- [Background] Al-Khateeb TH, Nusair Y. Effect of the proteolytic enzyme serrapeptase on swelling, pain and trismus after surgical extraction of mandibular third molars. Int J Oral Maxillofac Surg. 2008 Mar;37(3):264-8. doi: 10.1016/j.ijom.2007.11.011. Epub 2008 Feb 12. PMID 18272344
- [Background] Lokken P, Olsen I, Bruaset I, Norman-Pedersen K. Bilateral surgical removal of impacted lower third molar teeth as a model for drug evaluation: a test with ibuprofen. Eur J Clin Pharmacol. 1975 Apr 4;8(3-4):209-16. doi: 10.1007/BF00567117. PMID 786680
- [Background] Yamashita Y, Sano N, Shimohira D, Danjo A, Goto M. A parallel-group comparison study of celecoxib with loxoprofen sodium in third mandibular molar extraction patients. Int J Oral Maxillofac Surg. 2014 Dec;43(12):1509-13. doi: 10.1016/j.ijom.2014.09.002. Epub 2014 Sep 28. PMID 25270186
- [Background] Olmedo MV, Galvez R, Vallecillo M. Double-blind parallel comparison of multiple doses of ketorolac, ketoprofen and placebo administered orally to patients with postoperative dental pain. Pain. 2001 Feb 1;90(1-2):135-41. doi: 10.1016/s0304-3959(00)00396-1. PMID 11166979
- [Background] Wang D, He X, Wang Y, Li Z, Zhu Y, Sun C, Ye J, Jiang H, Cheng J. External root resorption of the second molar associated with mesially and horizontally impacted mandibular third molar: evidence from cone beam computed tomography. Clin Oral Investig. 2017 May;21(4):1335-1342. doi: 10.1007/s00784-016-1888-y. Epub 2016 Jun 18. PMID 27316639
- [Background] Ong CK, Lirk P, Tan JM, Sow BW. The analgesic efficacy of intravenous versus oral tramadol for preventing postoperative pain after third molar surgery. J Oral Maxillofac Surg. 2005 Aug;63(8):1162-8. doi: 10.1016/j.joms.2005.04.028. PMID 16094585
- [Background] Majid OW, Al-Mashhadani BA. Perioperative bromelain reduces pain and swelling and improves quality of life measures after mandibular third molar surgery: a randomized, double-blind, placebo-controlled clinical trial. J Oral Maxillofac Surg. 2014 Jun;72(6):1043-8. doi: 10.1016/j.joms.2013.12.035. Epub 2014 Jan 16. PMID 24589242
- [Background] Gaspani L, Limiroli E, Ferrario P, Bianchi M. In vivo and in vitro effects of bromelain on PGE(2) and SP concentrations in the inflammatory exudate in rats. Pharmacology. 2002 May;65(2):83-6. doi: 10.1159/000056191. PMID 11937778
- [Background] Bataineh AB, Batarseh RA. The effect of modified surgical flap design for removal of lower third molars on lingual nerve injury. Clin Oral Investig. 2017 Jul;21(6):2091-2099. doi: 10.1007/s00784-016-1999-5. Epub 2016 Nov 12. PMID 27837346
- [Background] Graziani F, D'Aiuto F, Gennai S, Petrini M, Nisi M, Cirigliano N, Landini L, Bruno RM, Taddei S, Ghiadoni L. Systemic Inflammation after Third Molar Removal: A Case-Control Study. J Dent Res. 2017 Dec;96(13):1505-1512. doi: 10.1177/0022034517722775. Epub 2017 Jul 31. PMID 28759304
- [Background] Mehra P, Reebye U, Nadershah M, Cottrell D. Efficacy of anti-inflammatory drugs in third molar surgery: a randomized clinical trial. Int J Oral Maxillofac Surg. 2013 Jul;42(7):835-42. doi: 10.1016/j.ijom.2013.02.017. Epub 2013 Mar 25. PMID 23535007
- [Background] Gallelli L. Escin: a review of its anti-edematous, anti-inflammatory, and venotonic properties. Drug Des Devel Ther. 2019 Sep 27;13:3425-3437. doi: 10.2147/DDDT.S207720. eCollection 2019. PMID 31631970
- [Background] Piecuch JF. What strategies are helpful in the operative management of third molars? J Oral Maxillofac Surg. 2012 Sep;70(9 Suppl 1):S25-32. doi: 10.1016/j.joms.2012.04.027. PMID 22916697
- [Background] Singhai A, Kambala R, Bhola N. Comparison of the efficacy of aescin and diclofenac sodium in the management of postoperative sequelae and their effect on salivary Prostaglandin E2 and serum C-reactive protein levels after surgical removal of impacted mandibular third molar: a randomized, double-blind, controlled clinical trial. F1000Res. 2024 Oct 30;13:106. doi: 10.12688/f1000research.145643.3. eCollection 2024. PMID 39507581
- [Background] Isola G, Matarese M, Ramaglia L, Iorio-Siciliano V, Cordasco G, Matarese G. Efficacy of a drug composed of herbal extracts on postoperative discomfort after surgical removal of impacted mandibular third molar: a randomized, triple-blind, controlled clinical trial. Clin Oral Investig. 2019 May;23(5):2443-2453. doi: 10.1007/s00784-018-2690-9. Epub 2018 Oct 11. PMID 30311061
- [Background] Sirtori CR. Aescin: pharmacology, pharmacokinetics and therapeutic profile. Pharmacol Res. 2001 Sep;44(3):183-93. doi: 10.1006/phrs.2001.0847. PMID 11529685